CLINICAL TRIAL: NCT05460000
Title: A Phase II Randomized, Open Label Non-inferiority Study of NiraParib Maintenance After 3 vs. 6 Cycles of Platinum-based Chemotherapy in completeLy debUlked Advanced HRDpositive High-grade Ovarian Cancer patientS in First Line Therapy (N-Plus)
Brief Title: A Phase II Randomized, Open Label Non-inferiority Study of NiraParib Maintenance After 3 vs. 6 Cycles of Platinum-based Chemotherapy in completeLy debUlked Advanced HRDpositive High-grade Ovarian Cancer patientS in First Line Therapy
Acronym: N-Plus
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: North Eastern German Society of Gynaecological Oncology (Other)
Collaborators: Institut für Klinische Krebsforschung IKF GmbH at Krankenhaus Nordwest (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NOGGO-ov53
Record Dates: First submitted 2022-07-07; First posted 2022-07-15 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Ovarian Cancer; Fallopian Tube Cancer; Primary Peritoneal Carcinoma; Clear Cell Carcinoma
Keywords: maintenance therapy; niraparib; HRDpositive; R0; primary tumor debulking; chemotherapy; LOH; carboplatin; paclitaxel; first line
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms; Adenocarcinoma, Clear Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Arm A (3 cycles of chemotherapy + maintenance therapy with niraparib) (Experimental): 3 cycles carboplatin + paclitaxel maintenance therapy with niraparib (starting dose 200 mg QD or 300 mg QD); maintenance continues until disease progression and/or death, unacceptable adverse event/s, patient and/or investigator decision, other protocol stopping criteria.
  Interventions: Drug: 3 cycles chemotherapy instead of 6 cycles chemotherapy
- Arm B (6 cycles of chemotherapy + maintenance therapy with niraparib) (Active Comparator): 6 cycles carboplatin + paclitaxel and maintenance therapy with niraparib (starting dose 200 mg QD or 300 mg QD); maintenance continues until disease progression and/or death, unacceptable adverse event/s, patient and/or investigator decision, other protocol stopping criteria.
  Interventions: Drug: 6 cycles chemotherapy

INTERVENTIONS:
Drug: 3 cycles chemotherapy instead of 6 cycles chemotherapy — We hypothesise that recurrence free survival in patients receiving 3 cycles of chemotherapy followed by maintenance with niraparib is not inferior to 6 cycles of chemotherapy followed by niraparib in advanced HRDpositive high-grade ovarian cancer patients with no residual tumor mass following primary tumor debulking.
  Arms: Arm A (3 cycles of chemotherapy + maintenance therapy with niraparib)
Drug: 6 cycles chemotherapy — Standard chemotherapy as comparator
  Arms: Arm B (6 cycles of chemotherapy + maintenance therapy with niraparib)

SUMMARY:
Multicenter, randomized, open label study including patients with advanced HRDpositive high-grade ovarian cancer, fallopian tube cancer, primary peritoneal cancer and clear cell carcinoma of the ovary with no residual tumor mass following primary tumor debulking to determine recurrence free survival in patients treated with 3 cycles carboplatin + paclitaxel and maintenance therapy with niraparib vs. 6 cycles carboplatin + paclitaxel and maintenance therapy with niraparib.

DETAILED DESCRIPTION:
This is a multicenter, randomized, open label study including patients with advanced (FIGO stage IIIA, IIIB, IIIC, or IV of the 2014 FIGO classification) HRDpositive high-grade ovarian cancer, fallopian tube cancer, primary peritoneal cancer and clear cell carcinoma of the ovary with no residual tumor mass following primary tumor debulking.

The main scope of the trial is to determine recurrence free survival in patients treated with 3 cycles carboplatin + paclitaxel and maintenance therapy with niraparib vs. 6 cycles carboplatin + paclitaxel and maintenance therapy with niraparib.

Patients will be randomized 1:1 to receive either 3 cycles carboplatin + paclitaxel maintenance therapy with niraparib (Arm A) or 6 cycles carboplatin + paclitaxel and maintenance therapy with niraparib (Arm B). Randomization will be performed according to the results of the NGS analysis and stratified either to BRCAm independent of LOH or LOHhigh/ BRCAwt, FIGO stage III vs. IV, and countries. In both of the arms, tumor assessments (CT or MRI) will be performed 9-12 weeks after the start of therapy (after 3rd cycle of chemotherapy), after another 9-12 weeks (during maintenance therapy in Arm A and after the 6th cycle of chemotherapy in Arm B) and every 6 months thereafter. The tumor marker CA-125 will be assessed every 12 weeks in both arms.

During chemotherapy treatment, clinical visits (blood cell counts, detection of toxicity) occur at least every 3 weeks (depending on the chemotherapy regimen). Serum pregnancy tests for WOCBP occur at least every 4 weeks. During maintenance therapy with niraparib, clinical visits (blood cell counts, detection of toxicity) occur every 4 weeks for the first 11 months and every 12 weeks thereafter. Serum pregnancy tests for WOCBP occur at least every 4 weeks. Complete physical examinations will take place every 12 weeks. Safety will be monitored continuously by careful monitoring of all adverse events (AEs) and serious adverse events (SAEs).

About 60 sites in 6 European countries will participate in this study to recruit 640 patients in 36 months.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent and obtained from the subject prior to performing any protocol-related procedures, including screening evaluations.
2. Female patient, age ≥ 18 years.
3. FIGO Stage III-IV high-grade ovarian cancer (all histological types, except mucinous histology)
4. Complete primary debulked patients (without any macroscopic residuals), confirmed by CT-Scan postoperatively.
5. Patients must have formalin-fixed, paraffin-embedded tumor samples available from the primary cancer for central NGS analysis and must be HRDpositive defined as BRCAmut independent of NOGGO GIS Score OR NOGGO GIS Score >83 independent of BRCA status, based on these results.
6. Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1.
7. Patients must be able to take oral medications.
8. Synchronous and secondary malignancies are allowed if the prognosis of the ovarian cancer is not affected. The investigator must contact the medical monitoring team before enrolling the patient in the clinical trial.
9. Patients must have normal organ and bone marrow function:

   1. Hemoglobin ≥ 10.0 g/dL independent of transfusion ≤ 14 days prior to screening hemoglobin assessment
   2. Absolute neutrophil count (ANC) ≥ 1.5 x 109/L
   3. Platelet count ≥ 100 x 109/L
   4. Total bilirubin ≤ 1.5 x institutional upper limit of normal (ULN); < 2 × ULN if hyperbilirubinemia is due to Gilbert's syndrome
   5. Aspartate aminotransferase /Serum Glutamic Oxaloacetic Transaminase (ASAT/SGOT)) and Alanine aminotransferase /Serum Glutamic Pyruvate Transaminase (ALAT/SGPT)) ≤ 2,5 x ULN
   6. Serum creatinine ≤ 1.5 x institutional ULN and creatinine clearance > 30 mL/min.
10. Postmenopausal or evidence of non-childbearing status for women of childbearing potential prior to the first dose of study treatment. Female patients of childbearing potential must have a negative serum pregnancy test result ≤3 days prior to administration of the first dose of study treatment.

Patients are considered to be of childbearing potential unless 1 of the following applies:

1. Considered to be permanently sterile. Permanent sterilization includes hysterectomy, bilateral salpingectomy, and/or bilateral oophorectomy; or
2. Is postmenopausal, defined as no menses for at least 12 months without an alternative medical cause. A high follicle-stimulating hormone (FSH) level consistently in the postmenopausal range (30 mIU/mL or higher) may be used to confirm a postmenopausal state in women not using hormonal contraception or hormonal replacement therapy; however, in the absence of 12 months of amenorrhea, a single FSH measurement is insufficient to confirm a postmenopausal state.

Female patients of reproductive potential must practice highly effective methods (failure rate < 1% per year) of contraception with their partners, if of reproductive potential, during treatment and for 6 months following the last dose of chemotherapy or the last dose of niraparib, whichever occurs later, or longer if requested by local authorities. Highly effective contraception includes: Ongoing use of progesterone only injectable or implantable contraceptives; Placement of an intrauterine device (IUD) or intrauterine system (IUS); Bilateral tubal occlusion; Sexual abstinence as defined as complete or true abstinence, acceptable only when it is the usual and preferred lifestyle of the patient; periodic abstinence (e.g., calendar, symptothermal, post-ovulation methods) is not acceptable; or Sterilization of the male partner, with appropriate post-vasectomy documentation of absence of sperm in ejaculate.

Exclusion Criteria:

1. Non-epithelial origin of the ovary, the fallopian tube or the peritoneum (i.e., germ cell tumors) and Ovarian tumors of low malignant potential (e.g., borderline tumors), or mucinous carcinoma of the ovary.
2. Low-grade ovarian, fallopian tube or peritoneal cancer.
3. Has known hypersensitivity to any of the study drugs or any of the excipients of any of the study drugs.
4. Has known hypersensitivity to platin-containing compounds other than carboplatin.
5. Patients posttransplant, including previous allogeneic bone marrow transplant.
6. Has undergone interval debulking of the tumor.
7. Has received any anti-cancer therapy for ovarian cancer other than primary surgery.
8. Administration of other simultaneous chemotherapy drugs, any other anti-cancer therapy or anti-neoplastic hormonal therapy, or simultaneous radiotherapy during the trial treatment period (hormonal replacement therapy is permitted as are steroidal antiemetics).
9. Has received prior treatment with a PARP inhibitor or has participated in a trial where any treatment arm included the administration of a PARP inhibitor.
10. Bevacizumab is planned to be given together with first line chemotherapy or as maintenance.
11. Clinically significant cardiovascular disease:

    1. Cerebrovascular accident or myocardial infarction or unstable angina ≤6 months before start of study treatment
    2. Severe cardiac arrhythmia (recent event or active or uncontrolled)
    3. New York Heart Association grade ≥2 congestive heart failure
    4. Uncontrolled hypertension (defined as systolic blood pressure >140 mmHg and/or diastolic blood pressure >90 mmHg), or history of hypertensive crisis, or hypertensive encephalopathy or posterior reversible encephalopathy syndrome
    5. History of stroke or transient ischemic attack ≤6 months before start of study treatment
    6. Coronary/peripheral artery bypass graft ≤6 months before start of study treatment
    7. Deep vein thrombosis or thromboembolic events ≤1 month before start of study treatment
12. History or evidence of brain metastases or spinal cord compression.
13. Known history of MDS or a pre-treatment cytogenetic testing result at risk for a diagnosis of MDS/AML.
14. Current, clinically relevant bowel obstruction at the time of randomization.
15. Patients with gastrointestinal disorders likely to interfere with absorption of the study medication.
16. Pregnant or lactating women, women of child-bearing potential who do not agree to the usage of highly effective contraception methods (see inclusion criteria) starting with the screening visit through at least 6 months after the last dose of chemotherapy treatment or through at least 1 month after the last dose of niraparib, whichever occurs later.
17. Participation in another clinical study with an investigational product immediately prior to randomization. Earliest time point for randomization is after the time required for the investigational product to undergo 5 half-lives has passed.
18. Has a known history of Human Immunodeficiency Virus (HIV) infection (known HIV1/HIV2 antibodies positive) or acquired immunodeficiency syndrome (AIDS) related illness.
19. Has a known history of Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus (defined as HCV RNA [qualitative] has been detected) infection.
20. Has active infection with SARS-CoV-2 (antigen test).
21. Has received a live vaccine or live-attenuated vaccine within 30 days prior to the first dose of chemotherapy treatment and while and 28 days after the last dose of trial treatment. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster, yellow fever, rabies, BCG, and typhoid vaccine. Administration of inactivated vaccines is allowed.
22. Patient has contraindications listed in the most recent SmPC.
23. Patient who might be dependent on the sponsor, CRO, site or the investigator.

22. In Germany: Patient who has been incarcerated or involuntarily institutionalized by court order or by the authorities § 40a S. 1 Nr. 2 AMG.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 640 (Estimated)
Dates: Start 2024-10-11 (Actual); Primary Completion 2032-10-01 (Estimated); Study Completion 2032-10-01 (Estimated)

PRIMARY OUTCOMES:
RFS | 8 years
  Recurrence free survival, defined as time from treatment randomization to the earliest date of assessment of first relapse or death by any cause

SECONDARY OUTCOMES:
Overall survival (OS) | 8 years
  time to event and rate at 3 and 5 years
TFST | 8 years
  Time to first subsequent treatment
TWIST (Time Without Symptoms of disease progression or Toxicity of treatment) | 8 years
  at baseline, 3, 6, and 12 months
PFS2 | 8 years
  Time from randomization until the date of second objective disease progression or death by any cause
Quality of Life (QoL) 1 | 8 years
  Patients are asked to answer the European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire Core 30 (QLQ-C30). Responses of questions 1-28 are based on a 4-point scale (1=not at all; 4=Very much), with a higher score indicating a high degree of symptomatology and must therefore be assessed negatively. Responses of questions 29 and 30 are based on a 7-point scale (1=Very poor; 7=Excellent), with a higher score indicating a better global health status.
Quality of Life 2 | 8 years
  Patients are asked to answer the EORTC QoL Questionnaire-Ovarian Cancer (QLQ-OV28). Responses are based on a 4-point scale (1=Not at all; 4=Very much), with a lower score indicating better symptoms.
Quality of Life/ Global health status 3 | 8 years
  Patients are asked to answer the short version of the SF-36 Health Survey (SF-12). The questionnaire contains a total of 12 questions with different response options. For questions 1, 8 and 12 there are 5 (1=excellent, 5=bad), for question 2-3 there are 3 (1=yes, very restricted, 3=no, not restricted at all) and for questions 9-11 there are 6 response options (1= always, 6 = never). Questions 4-7 can be answered with "Yes" or "No".
Safety Endpoints - safety of therapy (3 vs. 6 cycles of chemotherapy + niraparib maintenance therapy) according to CTCAE 5.0 criteria will be used as endpoint | 8 years
  The safety objective is to characterize the safety and tolerability of 3 vs. 6 cycles of chemotherapy followed by maintenance therapy with niraparib in advanced HRDpositive high-grade ovarian cancer patients with no residual tumor mass following primary tumor debulking. The following safety parameters will be analyzed: adverse events and serious adverse events graded per NCI CTCAE, Version 5.0 criteria with time to onset/recovery, causality and outcome; changes in laboratory values, vital signs since baseline, treatment discontinuations and reason for discontinuation, death and cause of death etc. concomitant medications will be collected with time and reasons of use. These are routine safety parameters collected and analyzed in Phase II /III oncology trials.
Cost effectiveness | 8 years
  The objective is to show that less cycles of chemotherapy are as efficient and at the same time less toxic. Additional cycles of chemotherapy significantly increase toxicity and therefore lead to an increase of costs regarding, e.g. in-patient treatment, concomitant medications to treat (S)AEs.

CONTACTS AND LOCATIONS:
Overall Officials: Jalid Sehouli, Prof. Dr. med., Principal Investigator — Lead coordinating investigator (LKP) according to AMG and representative of the sponsor
Locations (47):
- Universitätsklinik Innsbruck, Innsbruck, Austria
- Belgium (4):
  - Cliniques Universitaires St. Luc, Brussels
  - UZ Gent, Ghent
  - Jessa ziekenhuis, Hasselt
  - UZ Leuven, Leuven
- Czechia (3):
  - University Hospital Ostrava, Ostrava
  - General University Hospital in Prague, Prague
  - University Hospital Bulovka, Prague
- Germany (19):
  - Universitätsklinikum Aachen, Aachen
  - Klinikum Mittelbaden Baden-Baden Bühl, Baden-Baden
  - DRK-Kliniken Berlin-Köpenick, Berlin
  - Charité - Universitätsmedizin Berlin, Campus Virchow Klinikum, Berlin
  - ZAHO Bonn Onkologische Praxis, Bonn
  - Uniklinikum Bonn, Bonn
  - Klinikum Lippe, Detmold
  - Universitätsklinikum Carl Gustav Carus, Dresden
  - Florence-Nightingale-Krankenhaus Düsseldorf-Kaiserswerth, Düsseldorf
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - Universitätsklinik Göttingen, Göttingen
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - SLK-Kliniken Heilbronn, Heilbronn
  - Universitätsklinikum Schleswig-Holstein Campus Kiel, Kiel
  - Universitätsklinikum Leipzig, Leipzig
  - Universitätsklinik der Johannes-Gutenberg Universität Mainz, Mainz
  - Diakonie Klinikum Schwäbisch Hall, Schwäbisch Hall
  - Christliches Klinikum Unna Mitte, Unna
  - Helios Dr. Horst Schmidt Kliniken Wiesbaden, Wiesbaden
- Italy (10):
  - Policlinico St. Orsola Malpighi, Bologna
  - ASST Spedali Civili di Brescia, Brescia
  - ASST Lecco - Ospedale A. Manzoni, Lecco
  - IRCCS Istituto nazionale dei Tumori, Milan
  - AOU Cagliari, Monserrato
  - Istituto Oncologico Veneto (IOV), Padua
  - Azienda Ospedaliera Universitaria Pisana, Pisa
  - Azienda USL IRCCS Di Reggio Emilia, Reggio Emilia
  - AO Ordine Mauriziano, Torino
  - AOU Città della Salute e della Scienza di Torino - Ospedale Sant'Anna, Torino
- Spain (10):
  - Hospital General Universitario Dr. Balmis, Alicante
  - Hospital Virgen de las Nieves, Granada
  - Hospital Universitario Lucus Augusti, Lugo
  - CIOCC Clara Campal, Madrid
  - H. Althaia Manresa, Manresa
  - H.U. Virgen de la Macarena, Seville
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital Universitario Sant Joan de Reus, Tarragona
  - Hospital General Universitario de Valencia, Valencia
  - Hospital La Fe, Valencia

IPD SHARING:
Plan to Share IPD: Yes
Scientists may submit a request for scientific use of the data after the first publication. This request shall be examined by the working group and the leading PI. After signing an agreement, the anonymous data can be made available to the scientist (password protected).